CLINICAL TRIAL: NCT03173833
Title: Fulfilling Care Needs of Adolescents With Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 201612238RINA
Record Dates: First submitted 2017-05-24; First posted 2017-06-02 (Actual); Last update posted 2017-06-02 (Actual); Status verified 2017-04

CONDITIONS: Cancer
Keywords: cancer patients, quality of life
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Participants will not receive the outcome of their questionnaire in the form of computerized assessment with graphic outcome (CAGO) after the first time they fill in the questionnaire. And they will be able to discuss their care needs with their health care practitioners.
- Experimental group (Experimental): Participants will receive the outcome of their questionnaire in the form of computerized assessment with graphic outcome (CAGO) every time after the first time they fill in the questionnaire.
  And they will be able to discuss their care needs with their health care practitioners.
  Interventions: Other: CAGO questionnaire outcome

INTERVENTIONS:
Other: CAGO questionnaire outcome — Every time when cancer patients fulfill the following questionnaires, SDS, PTGI, CNS, PedsQL, the outcome of the questionnaires will be provided to the experimental group of the participants by using a computer assessment with graphic outcome.
  Other Names: computer assessment with graphic outcome (CAGO)
  Arms: Experimental group

SUMMARY:
The aim of phase 1 of this study is to develop a care need scale (CNS) for adolescents with cancer. The aim of phase 2 is to examine the mediating role of care needs between physical and psychosocial dysfunction and QoL, and to explore the recovery trajectory and its predictors regarding the care needs, physical and psychosocial factors, and the QoL of adolescents with cancer at the first, second, and third 3-month periods after initiating on-treatment and off-treatment. The aim of phase 3 is to examine the effectiveness of the computerized assessment with graphic outcome (CAGO) for fulfilling the care needs of adolescents with cancer, its acceptability for adolescents with cancer, and its usability for clinicians in pediatric oncology units.

ELIGIBILITY:
The inclusion criteria for adolescents with cancer are

1. 13-20 years of age
2. previously or currently treated for cancer
3. able to communicate in Chinese
4. able to comprehend the study information

Ages: 13 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 720 (Estimated)
Dates: Start 2017-08-01 (Estimated); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Symptom Distress Scale | 2 weeks
Beck Youth Inventories second edition | 2 weeks
Posttraumatic Growth Index | 2 weeks
Resilience Scale | 2 weeks
Care demand scale | 2 weeks
Pediatric Quality of Life | 2 weeks
Acceptability if E-scale | 2 weeks
Usability scale | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: SHIANN-TARNG LOU, Principal Investigator — National Taiwan University Hospital Department of Pediatrics
Locations (1):
- National Taiwan University Hospital, Test1, Test2, Taiwan

IPD SHARING:
Plan to Share IPD: No